CLINICAL TRIAL: NCT00923078
Title: Neurophysiological Targets for Cognitive Training in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: D7008-W
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2017-12-20 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Schizophrenia
Keywords: schizophrenia; cognitive remediation; rehabilitation; electrophysiology; neuropsychology
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Auditory-Visual Train Order (Experimental): 4 weeks (20 sessions) of auditory cognitive training (Brain Fitness) followed by 4 weeks (20 sessions) of visual cognitive training (Insight)
  Interventions: Behavioral: Auditory Cognitive Training; Behavioral: Visual Cognitive Training
- Visual-Auditory Train Order (Experimental): 4 weeks (20 sessions) of visual cognitive training (Insight) followed by 4 weeks (20 sessions) of auditory cognitive training (Brain Fitness)
  Interventions: Behavioral: Auditory Cognitive Training; Behavioral: Visual Cognitive Training

INTERVENTIONS:
Behavioral: Auditory Cognitive Training — The program entails six computer-based exercises that are designed to be very easy to use and require no computer experience. The exercises are calibrated to individual performance at the onset of training and adapt in difficulty to individual performance, giving constant feedback about progress. Each of the six exercises focuses on a distinct process: (1) auditory processing speed, (2) discriminating sounds, (3) sound precision, (4) sound sequencing, (5) working memory, and (6) narrative memory. Training was administered in a supervised clinical laboratory setting at a frequency of five 60-minute sessions per week over 4 weeks.
  Other Names: Brain Fitness by Posit Science
Behavioral: Visual Cognitive Training — The program entails five computer-based exercises that are designed to be very easy to use and require no computer experience. The exercises are calibrated to individual performance at the onset of training and, following our laboratory procedures, calibration testing is repeated every 5th session. Exercises adapt in difficulty to individual performance, giving constant feedback about progress. Each of the five exercises focuses on a distinct process: (1) visual precision, (2) visual processing speed, (3) divided attention, (4) visual working memory, and (5) useful field of view. Training was administered in a supervised clinical laboratory setting at a frequency of five 40-minute sessions per week over 4 weeks.
  Other Names: Cortex with Insight by Posit Science

SUMMARY:
The purpose of this study is to determine whether computer-based training of auditory and visual processing results in corresponding improvement in brain function in individuals with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is recognized as one of the leading causes of medical disability worldwide, ranked 9th overall by the World Health Organization, and affects more than 2 million Americans per year. There is considerable evidence to suggest that disability status in schizophrenia relates more directly to cognitive Impairment, involving attention, reasoning, and memory, than to characteristic symptoms of psychosis. Accordingly, the evaluation and advancement of interventions designed to restore cognitive function, generally termed cognitive remediation, is of critical importance to our rehabilitation mission. Recent randomized controlled trials of cognitive remediation in schizophrenia have found moderate gains in cognitive function and improved outcomes in important areas of community living. However, despite these encouraging findings, there remains sparse evidence in support of assumptions that (1) cognitive outcomes represent benefits of training-induced adaptive learning, (2) that training effects are specific to method of intervention, or (3) that change in cognitive test performance occurs through restoration of impaired neural circuitry in schizophrenia. This project will begin to address these issues by examining modality-specific effects of computer-based cognitive training on psychophysiological measures of sensory information processing. Training will be administered using two commercially available computer-based software packages, separately targeting auditory and visually-mediated processes using principles of bottom-up perceptual learning. Two psychophysiological paradigms, mismatch negativity (MMN) and P300 generation, will be administered as tests of early visual and auditory processing. MMN and P300 have been studied extensively in human neuroscience as probes of sensory echoic memory and attention engagement to contextually relevant information. Furthermore, reductions in MMN and P300 generation are reliably observed in schizophrenia, follow the course of a progressive neuropathological process, and correlate with severity of cognitive impairment. The specific aims of this study are to determine: (1) whether training selectively influences bottom-up (MMN) or top-down (P300) information processing, (2) whether training effects are modality (auditory vs. visual) specific, (3) whether baseline MMN and P300 predict, or rate-limit, training progress, and (4) whether pre-post change in cognitive test performance is mediated by neural-level change in MMN and P300 generation. Answers to these questions will provide information needed to structure cognitive training for maximum benefit in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia or schizoaffective disorder
* Age between 18 & 70
* minimum of 30 days since discharge from last hospitalization
* minimum of 30 days since last change in psychiatric medications
* receiving mental health services
* no housing changes in the past 30 days

Exclusion Criteria:

* current diagnosis of alcohol or substance abuse
* history of brain trauma or neurological disease
* chart diagnosis of mental retardation or premorbid intelligence < 70 based on Wechsler Test of Adult Reading (WTAR) full-scale estimated IQ
* auditory or visual impairment that would interfere with study procedures

  * a sample of 20 healthy community volunteers was also recruited according to these criteria and tested, without intervention, as a normative reference sample for MMN and P300 measures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason K Johannesen, PhD, Principal Investigator — VA Connecticut Health Care System (West Haven)
Locations (1):
- VA Connecticut Health Care System (West Haven), West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Healthy comparison subjects completed a single assessment at baseline and did not receive intervention or follow-up testing.
Groups:
- Auditory Then Visual Cognitive Training: 20 individuals with schizophrenia randomized to 4 weeks (20 sessions) of auditory training (Brain Fitness) followed by 4 weeks (20 sessions) of visual training (Insight).
- Visual Then Auditory Cognitive Training: 20 individuals with schizophrenia randomized to 4 weeks (20 sessions) of visual training (Insight) followed by 4 weeks (20 sessions) of auditory training (Brain Fitness).
- Healthy Comparison: A sample healthy community volunteers participated in a single test session to provide normative comparison data on neurophysiological (P300, MMN) outcome measures
Period: First Intervention (Weeks 1-4)
Arm/Group | Auditory Then Visual Cognitive Training | Visual Then Auditory Cognitive Training | Healthy Comparison
Started | 20 | 20 | 20
Completed | 19 | 19 | 0
Not Completed | 1 | 1 | 20
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — No intervention per protocol | 0 | 0 | 20
Period: Second Intervention (Weeks 5-8)
Arm/Group | Auditory Then Visual Cognitive Training | Visual Then Auditory Cognitive Training | Healthy Comparison
Started | 19 | 19 | 0 (Healthy Comparison sample subjects completed only a single test session (baseline))
Completed | 19 | 19 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Auditory-Visual Train Order: N = 20 participants with schizophrenia randomized to 4 weeks (20 sessions) of auditory training (Brain Fitness) followed by 4 weeks (20 sessions) of visual training (Insight)
- Visual-Auditory Train Order: N = 20 participants with schizophrenia randomized to 4 weeks (20 sessions) of visual training (Insight) followed by 4 weeks (20 sessions) of auditory training (Brain Fitness)
- Healthy Comparison: N = 20 healthy community volunteers participated in a single test session to provide normative comparison data
- Total: Total of all reporting groups
Arm/Group | Auditory-Visual Train Order | Visual-Auditory Train Order | Healthy Comparison | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 20 | 58
  >=65 years | 1 | 1 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.65 (12.26) | 46.55 (12.85) | 39.15 (13.39) | 43.78 (13.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 9 | 26
  Male | 13 | 10 | 11 | 34
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60
IQ [Mean (Standard Deviation); unit: units on a scale] — Estimated IQ derived from age, gender, race normative performance of the Wechsler Test of Adult Reading (WTAR). IQ scores reported in standard form with M = 100, SD = 15
  units on a scale | 95.20 (14.83) | 87.70 (12.32) | 103.26 (13.86) | 95.25 (14.90)
Cognitive Composite Score [Mean (Standard Deviation); unit: t-score] — MATRICS Consensus Cognitive Battery (MCCB) cognitive composite score, reported as age- and gender-corrected t-score (M=50, SD =10) with higher score indicating better cognitive ability
  t-score | 36.35 (12.86) | 30.40 (12.87) | 45.95 (13.70) | 37.57 (14.45)
Positive and Negative Syndrome Scale (PANSS) [Mean (Standard Deviation); unit: units on a scale] — Clinical interview rating of schizophrenia symptom severity. The PANSS has a possible score range of 30-210 across 30 items, with higher scores indicating greater symptom distress. Per test literature, stable outpatients typically score between 60-80, and inpatient cases seldom exceed 80-150 at highest severity. Population: The PANSS is a schizophrenia symptom severity measure, ratings not obtained in healthy community sample
  units on a scale
    number analyzed (Participants) | 20 | 20 | 0 | 40
    (all) | 56.8 (12.89) | 56.8 (13.94) |  | 56.8 (13.25)

OUTCOME MEASURES:

1. Primary Outcome: Visual Target Detection (P300 Event-related Potential Amplitude) Change
Description: Visual P300 was measured in a 3-stimulus target detection task with target stimuli (10%; large circle) presented in pseudo random order amidst a series of novel (10%; fractal), and standard (80%; small circle) images on a 24" LCD monitor at 100cm viewing distance. Subjects are instructed to press a reaction time button with the preferred hand to Targets only, giving equal importance to speed and accuracy. Primary analysis are based on Target "P300b" identified as the most positive amplitude deflection within the window of 250-550ms post stimulus at posterior midline electrode Pz. The P300b component is thought to reflect cognitive processes involved in memory updating and decision making. P300 reported as difference scores from baseline with negative values indicating increased P300.
Time Frame: Baseline; Post 4 weeks (treatment crossover); Post 8 weeks
Measure: Mean (Standard Error); unit: microvolts (uV)
Groups:
- Auditory Cognitive Training: 4 weeks (20 sessions) of auditory cognitive training (Brain Fitness) completed either before or following 4 weeks (20 sessions) of visual cognitive training (Insight)
- Visual Cognitive Training: 4 weeks (20 sessions) of visual cognitive training (Insight) completed either before or following 4 weeks (20 sessions) of auditory cognitive training (Brain Fitness)
Arm/Group | Auditory Cognitive Training | Visual Cognitive Training
Number analyzed (Participants) | 38 | 38
microvolts (uV) | 2.20 (1.02) | -0.72 (1.02)
Statistical Analysis 1: Comparison: Auditory Cognitive Training; Null hypothesis is that there is no difference between baseline and post-training scores. Linear mixed models tested fixed effects of period (3 levels; baseline, post 4-weeks, post 8 weeks), condition (3 levels; baseline, Auditory Cognitive Training, Visual Cognitive Training) and the period x condition interaction. Final model parameters were selected according to Bayesian Information Criteria. Alpha=.05 (2-sided); Test type: Other; p < 0.05, Mixed Models Analysis; Mean Difference (Net) = 2.20, 95% CI 2-sided [0.17 to 4.23], Standard Error of Mean 1.02 — contrast calculated as baseline minus Auditory Training
Statistical Analysis 2: Comparison: Visual Cognitive Training; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.48, Mixed Models Analysis; Mean Difference (Net) = -0.72, 95% CI 2-sided [-2.75 to 1.31], Standard Error of Mean 1.02 — contrast calculated as baseline minus Visual Training
Statistical Analysis 3: Comparison: Auditory Cognitive Training vs Visual Cognitive Training; Null hypothesis is that there is no difference between post-training scores in Auditory vs. Visual Cognitive Training conditions. Linear mixed models tested fixed effects of period (3 levels; baseline, post 4-weeks, post 8 weeks), condition (3 levels; baseline, Auditory Cognitive Training, Visual Cognitive Training) and the period x condition interaction. Final model parameters were selected according to Bayesian Information Criteria. Alpha=.05 (2-sided); Test type: Superiority or Other; p < 0.01, Mixed Models Analysis; Mean Difference (Final Values) = -2.92, 95% CI 2-sided [-4.95 to -0.90], Standard Error of Mean 1.02 — contrast calculated as Auditory Training minus Visual Training

2. Primary Outcome: Auditory Mismatch Negativity (MMN) Amplitude Change
Description: Auditory MMN is a fronto-central, mid-latency, potential generated by the auditory cortex in response to deviation in a repetitive stimulus sequence. MMN was assessed using a 3-deviant paradigm in which a series of standard tones (633 Hz, 50ms duration,90%) is interrupted by deviants (10%) that differ either by (1) pitch (1000Hz, 50ms), (2) duration (633 Hz, 100ms), or (3) both (1000Hz, 100ms). MMN was tested concurrently with Visual P300 using a combined task in which subjects were instructed to ignore the auditory stimuli and focus on the visual stimuli. MMN is scored by subtracting each deviant ERP waveform from the standard waveform and measuring the most negative deflection in a window of 50 to 265ms post-stimulus from the resulting difference wave. Primary analysis is based on the combined deviant condition scored at the frontal midline (Fz) electrode site. MMN reported as difference scores from baseline with positive values indicating increased MMN.
Time Frame: Baseline; Post 4 weeks (treatment crossover); Post 8 weeks
Measure: Mean (Standard Error); unit: microvolts (uV)
Arm/Group | Auditory Cognitive Training | Visual Cognitive Training
Number analyzed (Participants) | 38 | 38
microvolts (uV) | 0.67 (0.29) | 0.51 (0.29)
Statistical Analysis 1: Comparison: Auditory Cognitive Training; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Mean Difference (Net) = 0.67, 95% CI 2-sided [0.08 to 1.25], Standard Error of Mean .295 — contrast calculated as baseline minus Auditory Training
Statistical Analysis 2: Comparison: Visual Cognitive Training; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.09, Mixed Models Analysis; Mean Difference (Net) = .51, 95% CI 2-sided [-0.08 to 1.09], Standard Error of Mean .295 — contrast calculated as baseline minus Visual Training
Statistical Analysis 3: Comparison: Auditory Cognitive Training vs Visual Cognitive Training; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.59, Mixed Models Analysis; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.75 to 0.43], Standard Error of Mean .295 — contrast calculated as Auditory Training minus Visual Training

3. Primary Outcome: MCCB Cognitive Composite Score Change
Description: The Cognitive Composite score is derived from the MATRICS Consensus Cognitive Battery (MCCB). The MCCB consists of 10 tests and provides standard scores for each according to seven cognitive domains: (1) speed of processing, (2) attention/vigilance, (3) working memory (verbal and visual), (4) verbal learning, (5) visual learning, (6) reasoning and problem solving, and (7) social cognition. The primary dependent measures derived from the MCCB for purpose of this study is the cognitive composite score, computed as the average of standard (t-scores) scores from each domain excluding social cognition. MCCB Composite reported as difference scores from baseline with negative values indicating higher test performance.
Time Frame: Baseline; Post 4 weeks (treatment crossover); Post 8 weeks
Population: Of N=40 randomized, analysis was based on 38 who completed intervention and post-testing. Across conditions, participants completed, on average, 14.61 hrs of training in Period 1 (12.53 visual, 16.70 auditory) and 14.41 hrs in Period 2 (13.00 visual, 15.92 auditory)
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Auditory Cognitive Training | Visual Cognitive Training
Number analyzed (Participants) | 38 | 38
t-score | -2.03 (0.75) | -2.45 (0.75)
Statistical Analysis 1: Comparison: Auditory Cognitive Training; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis — Post-test scores following Auditory Cognitive Training as compared to baseline, tested at alpha = 0.05 (uncorrected); Mean Difference (Net) = -2.03, 95% CI 2-sided [-3.53 to -0.52], Standard Error of Mean 0.75 — contrast calculated as baseline minus Auditory Training
Statistical Analysis 2: Comparison: Visual Cognitive Training; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis — Post-test scores following Visual Cognitive Training as compared to baseline, tested at alpha = 0.05 (uncorrected); Mean Difference (Net) = -2.45, 95% CI 2-sided [-3.95 to -0.94], Standard Error of Mean 0.75 — contrast calculated as baseline minus Visual Training
Statistical Analysis 3: Comparison: Auditory Cognitive Training vs Visual Cognitive Training; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.58, Mixed Models Analysis — Post-test scores following Auditory Cognitive Training as compared to Visual Cognitive Training, tested at alpha = 0.05 (uncorrected); Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-1.93 to 1.08], Standard Error of Mean 0.75 — contrast calculated as Auditory Training minus Visual Training

4. Secondary Outcome: Visual Learning (BVMT-R) Change
Description: The visual learning domain of the MCCB is assessed using the Brief Visuospatial Memory Test-Revised (BVMT-R). In three Learning Trials, the respondent views a stimulus display for 10 seconds and is then asked to draw as many of the figures as possible in their correct location on a page in the response booklet. Scores represent overall accuracy across the three trials, with higher scores indicating better learning. Analysis is based on age- and gender-corrected t-scores. BVMT-R reported as difference scores from baseline with negative values indicating higher test performance.
Time Frame: Baseline; Post 4 weeks (treatment crossover); Post 8 weeks
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Auditory Cognitive Training | Visual Cognitive Training
Number analyzed (Participants) | 38 | 38
t-score | -2.92 (1.55) | -3.24 (1.55)
Statistical Analysis 1: Comparison: Auditory Cognitive Training; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.06, Mixed Models Analysis; Mean Difference (Net) = -2.92, 95% CI 2-sided [-6.02 to 0.18], Standard Error of Mean 1.55 — contrast calculated as baseline minus Auditory Training
Statistical Analysis 2: Comparison: Visual Cognitive Training; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Mean Difference (Net) = -3.24, 95% CI 2-sided [-6.34 to -0.14], Standard Error of Mean 1.55 — contrast calculated as baseline minus Visual Training
Statistical Analysis 3: Comparison: Auditory Cognitive Training vs Visual Cognitive Training; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.84, Mixed Models Analysis; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-3.42 to 2.78], Standard Error of Mean 1.55 — contrast calculated as Auditory Training minus Visual Training

5. Secondary Outcome: Verbal Learning (HVLT-R) Change
Description: The verbal learning domain of the MCCB is assessed using the Hopkins Verbal Learning Test-Revised (HVLT-R). In three Learning Trials, the respondent listens to a 12-item word list read by an examiner and is then asked to recall as many of the words as possible from memory. Scores represent overall accuracy across the three trials, with higher scores indicating better learning. Analysis is based on age- and gender-corrected t-scores. HVLT-R reported as difference scores from baseline with negative values indicating higher test performance.
Time Frame: Baseline; Post 4 weeks (treatment crossover); Post 8 weeks
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Auditory Cognitive Training | Visual Cognitive Training
Number analyzed (Participants) | 38 | 38
t-score | 0.62 (1.04) | 0.03 (1.03)
Statistical Analysis 1: Comparison: Auditory Cognitive Training; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.55, Mixed Models Analysis; Mean Difference (Net) = 0.62, 95% CI 2-sided [-1.45 to 2.69], Standard Error of Mean 1.04 — contrast calculated as baseline minus Auditory Training
Statistical Analysis 2: Comparison: Visual Cognitive Training; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.98, Mixed Models Analysis; Mean Difference (Net) = 0.03, 95% CI 2-sided [-2.02 to 2.07], Standard Error of Mean 1.03 — contrast calculated as baseline minus Visual Training
Statistical Analysis 3: Comparison: Auditory Cognitive Training vs Visual Cognitive Training; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.57, Mixed Models Analysis; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-2.66 to 1.47], Standard Error of Mean 1.04 — contrast calculated as Auditory Training minus Visual Training

6. Secondary Outcome: Visual Working Memory (Spatial Span) Change
Description: Visual working memory is assessed in the MCCB using the Spatial Span task of the Wechsler Memory Scales-III. Using a board on which 10 cubes are irregularly spaced, the examiner taps patterns of increasing length. The respondent is asked to follow by tapping the pattern in the same or reverse sequence. Scores represent total accuracy combined over forward and reverse span conditions. Analysis is based on age- and gender-corrected t-scores. Spatial Span reported as difference scores from baseline with negative values indicating higher test performance.
Time Frame: Baseline; Post 4 weeks (treatment crossover); Post 8 weeks
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Auditory Cognitive Training | Visual Cognitive Training
Number analyzed (Participants) | 38 | 38
t-score | -0.60 (1.27) | -0.92 (1.27)
Statistical Analysis 1: Comparison: Auditory Cognitive Training; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.63, Mixed Models Analysis; Mean Difference (Net) = -0.60, 95% CI 2-sided [-3.14 to 1.93], Standard Error of Mean 1.27 — contrast calculated as baseline minus Auditory Training
Statistical Analysis 2: Comparison: Visual Cognitive Training; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.47, Mixed Models Analysis; Mean Difference (Net) = -0.92, 95% CI 2-sided [-3.45 to 1.61], Standard Error of Mean 1.27 — contrast calculated as baseline minus Visual Training
Statistical Analysis 3: Comparison: Auditory Cognitive Training vs Visual Cognitive Training; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.80, Mixed Models Analysis; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-2.85 to 2.22], Standard Error of Mean 1.27 — contrast calculated as Auditory Training minus Visual Training

7. Secondary Outcome: Auditory Working Memory (LNS) Change
Description: Auditory working memory is assessed in the MCCB using the Letter-Number Sequencing (LNS) task. LNS is an orally administered test in which and examiner reads strings of numbers and letters, of increasing length over trials, and the respondent mentally reorders the string and reports back to the examiner verbally. Scores represent total number of accurate trials. Analysis is based on age- and gender-corrected t-scores. LNS reported as difference scores from baseline with negative values indicating higher test performance.
Time Frame: Baseline; Post 4 weeks (treatment crossover); Post 8 weeks
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Auditory Cognitive Training | Visual Cognitive Training
Number analyzed (Participants) | 38 | 38
t-score | -1.10 (0.98) | -1.47 (0.97)
Statistical Analysis 1: Comparison: Auditory Cognitive Training; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.26, Mixed Models Analysis; Mean Difference (Net) = -1.10, 95% CI 2-sided [-3.06 to 0.85], Standard Error of Mean 0.98 — contrast calculated as baseline minus Auditory Training
Statistical Analysis 2: Comparison: Visual Cognitive Training; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.13, Mixed Models Analysis; Mean Difference (Net) = -1.47, 95% CI 2-sided [-3.41 to 0.46], Standard Error of Mean 0.97 — contrast calculated as baseline minus Visual Training
Statistical Analysis 3: Comparison: Auditory Cognitive Training vs Visual Cognitive Training; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.71, Mixed Models Analysis; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-2.32 to 1.58], Standard Error of Mean 0.98 — contrast calculated as Auditory Training minus Visual Training

ADVERSE EVENTS:
Time Frame: Events were monitored during the active study period of 60 days
Groups:
- Auditory Cognitive Training: Individuals with schizophrenia randomized to 4 weeks (20 sessions) of auditory training (Brain Fitness)
- Visual Cognitive Training: Individuals with schizophrenia randomized to 4 weeks (20 sessions) of visual training (Insight)
Arm/Group | Auditory Cognitive Training | Visual Cognitive Training | Healthy Comparison
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/20
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes